CLINICAL TRIAL: NCT07201064
Title: An Exploratory Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of SZ1003 Injection in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of SZ1003 Injection in Patients With Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong ProCapZoom Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLKR-SZ1003-I-101
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Intervention Model Description: multiple Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SZ1003 injection (Experimental): once every two weeks at a dose of SZ1003 injection per infusion
  Interventions: Drug: SZ1003 injection

INTERVENTIONS:
Drug: SZ1003 injection — once every two weeks at a dose of SZ1003 injection per infusion.
  Other Names: SZ1003

SUMMARY:
This study is a "3+3" dose-escalation, open-label, multiple-dose clinical trial.

DETAILED DESCRIPTION:
This study is a "3+3" dose-escalation, open-label, multiple-dose clinical trial. To evaluate the safety, tolerability, and preliminary efficacy of SZ1003 injection in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old, including the boundary value, no gender restriction;
* Meet the diagnostic criteria for advanced hepatocellular carcinoma established by histopathology and/or cytology, and have experienced failure of second-line therapy for advanced HCC (per 2024 CSCO Guidelines for Primary Liver Cancer). Patients must have progressed during or after at least two prior lines of standard systemic therapy (intolerant or refractory), with radiologically documented disease progression. Eligible stages are Barcelona Clinic Liver Cancer stage B or C, or stage IIb/IIIa/IIIb as defined in the 2024 Chinese Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (stage-IIb patients must be deemed unsuitable for surgery or TACE);
* Have at least one measurable or evaluable lesion per RECIST 1.1;
* GPC3 positivity confirmed by immunohistochemistry on a clinical pathology section;
* Child-Pugh classification: class A or class B (≤ 7 points) (See Appendix 1 for the Child-Pugh classification table).;
* ECOG performance status: the score is 0 or 1 (See Appendix 2 for the ECOG-PS scoring table);
* Renal function: serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min by Cockcroft-Gault;
* Coagulation: INR, APTT, and PT ≤ 1.5 × ULN without anticoagulant therapy.
* Able to undergo routine peripheral venous blood collection, establish adequate venous access, and have no contraindications to peripheral blood procurement.
* Women of child-bearing potential must have a negative serum or urine pregnancy test within 14 days before enrollment and agree to use effective non-hormonal contraception (e.g., condoms, non-medicated IUD) throughout the trial to minimize the risk of pregnancy. Men with partners of child-bearing potential and women of child-bearing potential must maintain effective contraception from screening until 12 months after the last cell infusion.
* Willing to participate in the study, fully informed of the study and sign the informed consent form; willing to comply with all trial procedures.

Exclusion Criteria:

* Patients who have previously undergone liver transplantation, organ allotransplantation, allogeneic stem-cell transplantation, and renal-replacement therapy.
* Clinically detectable hepatic encephalopathy or those requiring pharmacological treatment for hepatic encephalopathy.
* Moderate-to-severe ascites attributable to portal hypertension or cirrhosis.
* History of leptomeningeal or central-nervous-system metastases.
* Neurologic disorder ≥ Grade 2 (CTCAE).
* Having experienced esophageal or gastric variceal bleeding due to portal hypertension within the past 3 months. Patients with evidence of portal hypertension and a high bleeding risk as assessed by the investigator.
* Having experienced any life-threatening bleeding events within the past 3 months, including those requiring transfusion, surgery, local treatment, or continuous pharmacological therapy.
* History of stroke or central nervous system hemorrhage; Prior stroke, CNS hemorrhage, TIA, or RIND within 6 months.
* Uncontrolled hypertension (SBP > 140 mmHg or DBP > 90 mmHg despite optimal therapy), hypertensive crisis, or hypertensive encephalopathy.
* Symptomatic CHF (NYHA ClassII-IV), Symptomatic or poorly controlled arrhythmias. Electrocardiogram (ECG) showing clinically significant abnormalities, or QTc interval ≥ 450 milliseconds in men, ≥ 470 milliseconds in women (≥ 480 milliseconds for subjects with bundle branch block on consecutive ECGs) (calculated using Fridericia's formula).
* Severe bleeding diathesis, coagulopathy, or ongoing thrombolytic therapy.
* A history of or current pulmonary fibrosis, interstitial pneumonitis, pneumoconiosis, drug-related pneumonitis, or severely impaired pulmonary function.
* HBsAg-positive subjects with HBV-DNA above the lower limit of detection at the study site must receive at least 7 days of antiviral therapy before the first dose and are willing to continue antiviral treatment for hepatitis B as required during the study to be eligible for enrollment. HBsAg-negative but HBcAb-positive subjects with HBV-DNA below the lower limit of detection at the study site will be closely monitored for HBV-DNA and liver transaminase levels during the dosing period. If HBV reactivation occurs during the treatment period, these subjects must agree to immediately initiate antiviral therapy for hepatitis B to remain eligible. All such subjects must be willing to continue antiviral treatment for hepatitis B for at least 6 months after the last dose, and the investigator may follow up on hepatitis B markers based on individual patient circumstances. Active hepatitis C: HCV antibody-positive with HCV-RNA levels above the lower limit of detection at the study site; co-infection with hepatitis B and hepatitis C.
* Active tuberculosis (TB), subjects currently receiving anti-TB treatment or those who have received anti-TB treatment within 1 year before the first dose.
* HIV-positive or active syphilis.
* Subjects with active or poorly controlled serious infections; those who have had severe infections within 4 weeks before peripheral blood collection, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications.
* Active autoimmune disease requiring systemic therapy (immunosuppressants, corticosteroids, or DMARDs) within 2 years and not adequately controlled.
* History of malignancy (other than HCC) within 5 years.
* Known hypersensitivity to study drug or its components.
* Pregnant or lactating women.
* Subjects deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | from subjects receiving administration to Week 24 post-administration
  Incidence and severity of adverse events from subjects receiving administration to Week 24 post-administration.
Serious adverse events | from subjects receiving administration to Week 24 post-administration
  Incidence and severity of adverse events from subjects receiving administration to Week 24 post-administration.

SECONDARY OUTCOMES:
Objective Response Rate | from subjects receiving administration to Week 24 post-administration
  Every 8 weeks, objective response rate will be assessed according to RECIST 1.1..
Disease Control Rate | from subjects receiving administration to Week 24 post-administration
  Every 8 weeks, disease control rate will be assessed according to RECIST 1.1..
Duration of Response | from subjects receiving administration to Week 24 post-administration
  Every 8 weeks, duration of response will be assessed according to RECIST 1.1..
Progression-Free Survival | from subjects receiving administration to Week 24 post-administration
  Every 8 weeks, progression-free survival will be assessed according to RECIST 1.1..
Overall Survival | from subjects receiving administration to Week 24 post-administration
  Every 8 weeks, overall survival will be assessed according to RECIST 1.1..

IPD SHARING:
Plan to Share IPD: No